CLINICAL TRIAL: NCT04486768
Title: Orphan Disease Center CDKL5 Deficiency Disorder International Patient Registry
Brief Title: International CDKL5 Registry
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Loulou Foundation (Other); International Foundation for CDKL5 Research (Unknown); CDKL5 Alliance (Unknown)
Responsible Party: Sponsor
Other Study IDs: ODC-IPR-CDD-01
Record Dates: First submitted 2020-02-06; First posted 2020-07-27 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: CDKL5 Deficiency Disorder (CDD)
Keywords: CDKL5; CDD; CDKL5 Disorder; CDKL5 Deficiency; pediatric epilepsy; epilepsy; CDKL5 Registry; CDKL5 Patient Registry; CDD Registry; CDD Patient Registry
MeSH Terms: conditions — CDKL5 deficiency disorder; Epilepsies, Myoclonic; Epilepsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey Instrument — This registry contains several surveys that will be released for patient/caregiver completion at enrollment and at time points following enrollment. These surveys can be completed on any computer that is connected to the internet.

SUMMARY:
Owing to the recent classification of CDKL5 Deficiency Disorder (CDD) as a unique disorder, there is a limited understanding of overall disease natural history and meaningful outcome measures. An international patient registry aimed at collecting both patient/caregiver and clinician-entered demographic, patient-reported outcome (PRO) and treatment data would benefit both the scientific and patient communities. This CDD registry will follow up to 500 patients diagnosed with CDD over several years through both the patients/caregivers and their clinicians. Initial data will be collected upon enrollment in the registry, followed by the collection of additional CDD-specific data on a bi-annual/ annual basis. No procedures will be performed as part of this registry. Clinician-entered data will be collected following standard of care visits conducted as part of patients' ongoing clinical care. Ultimately, the goal is to create a contact registry to allow patients/families to be alerted about relevant clinical trials and to collect valuable information that is accessible to the patient and scientific communities, thereby aiding and encouraging research in CDD.

ELIGIBILITY:
Inclusion Criteria:

* Person of any age, living or deceased;
* Be a patient or the legal guardian (parent or caregiver) of a patient with a diagnosis of CDD (Diagnoses must be confirmed by a clinician or genetic test);
* Have the ability to understand and complete an informed consent process where applicable per local regulations or have a legal guardian to provide consent on the patient's behalf if the patient is under the legal age, per local regulations, or otherwise unable to provide consent.

Exclusion Criteria:

* Patient with a diagnosis of CDD who is under the legal age, per local regulations, enrolling without a legal guardian;
* Legal guardian of a patient who is 1) over the legal age, per local regulations, and 2) is able to read and provide consent and enter data. (We require that patients over the legal age who are capable of reading and understanding and informed consent provide data directly.)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: We expect to enroll up to 500 CDD patients over a 5 year period. As CDD affects people globally, we anticipate enrollment from several countries. Patients will learn about the registry through the Orphan Disease Center's social media presence, disease-specific foundations, other families impacted by CDD and/or physicians involved in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of different mutation types and genotype-phenotype correlations in CDKL5 Deficiency Disorder (CDD). | 1 year
  Measured by data obtained from genetic reports of enrolled patients.
Caregiver reported longitudinal assessments to quantify seizure frequency over time. | 1 year
  Measured by the mean number of seizures reported at 1 week intervals over a 1 year period.
Caregiver reported longitudinal assessment of sleep quality in patients over time. | up to 5 years
  Measured by mean rating of sleep disruptions indicated by collective score of night terrors and excessive daytime somnolence at 1 year intervals over a period of 5 years.
Caregiver reported assessment of GI disturbances in patients over time and across age groups. | up to 5 years
  Measured by rating of gastroesophageal reflux, dysphagia, constipation, bowel incontinence, bloating and distension at 1 year intervals over a period of 5 years.
Caregiver reported longitudinal assessment of supplement use for the treatment of CDKL5 Deficiency Disorder (CDD) as an adjunct to prescription medications. | up to 5 years
  Measured by percent of patients using clinician prescribed or over the counter (OTC) supplements.
Caregiver reported longitudinal assessment of diet use for the treatment of CDKL5 Deficiency Disorder (CDD) as an adjunct to prescribed medications. | up to 5 years
  Measured by percent of subjects using clinician prescribed or self-selected diets e.g Ketogenic diet.

SECONDARY OUTCOMES:
Caregiver reported time to attainment of developmental milestones. | up to 5 years
  Measured by rating of indicated skills (e.g. sitting up, crawling, standing, hand use and gestures) at 1 year intervals over a period of 5 years.
Medication use in patients by age group. | 1 year
  Measured by percentage of patients reporting use of selected approved prescription medications as part of CDKL5 Deficiency Disorder (CDD) management plan.
Frequency of hospitalization in CDKL5 Deficiency Disorder (CDD) patients. | up to 5 years
  Measured by the mean number of hospital visits leading to admissions at 1 year intervals over 5 years.
Frequency of respiratory infections in CDKL5 Deficiency Disorder (CDD) patients. | up to 5 years
  Measured by the percentage of patients reporting a respiratory infection at 1 year intervals over 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Lavery, PhD, Principal Investigator — Director, CDKL5 Program of Excellence, Orphan Disease Center
Locations (1):
- University of Pennsylvania Orphan Disease Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available by request to the Orphan Disease Center Data Access Board (DAB).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available beginning 1 year after study enrollment target reached.
Access Criteria: Researchers studying CDKL5 Deficiency Disorder, epilepsy, and related rare diseases.
URL: https://www.cdkl5registry.org